CLINICAL TRIAL: NCT05241977
Title: MINIMUM EFFECTIVE AND MAXIMUM DIAPHRAGM-SPARING VOLUME OF BUPIVACAİNE FOR ULTRASOUND GUIDED ANTERIOR SUPRASCAPULAR NERVE BLOCK
Brief Title: MINIMUM EFFECTIVE VOLUME OF BUPIVACAİNE FOR ANTERIOR SUPRASCAPULAR NERVE BLOCK
Status: Completed | Type: Observational
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Sami Kaan Coşarcan, MD, V.K.V. American Hospital, Istanbul
Other Study IDs: Cosarcan1
Record Dates: First submitted 2022-02-07; First posted 2022-02-16 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Shoulder Pain; Supraspinatus Tendinitis; Bankart Lesions
Keywords: regional anesthesia; shoulder arthroscopy; ortopaedic anesthesia; brachial plexus blocks; diaphragm sparing nerve blocks
MeSH Terms: conditions — Shoulder Pain; Bankart Lesions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Anterior suprasscapular nerve block: A single researcher will perform the nerve blocks of all participants.
  Interventions: Procedure: anterior supra scapular nerve block

INTERVENTIONS:
Procedure: anterior supra scapular nerve block — nerve block for postoperative pain

SUMMARY:
Various local anesthetic volumes are used in the literature for anterior suprascapular nerve block (ASSB). There are different studies between 15 ml and 5 ml. Effective local anesthetic volume studies for ASSB have not yet been performed. Our study is aimed to investigate the minimum effective local anesthetic volume for ASSB.

DETAILED DESCRIPTION:
Peripheral nerve blockade reduces pain scores and opioid consumption and increases patient satisfaction within the first 24 h after shoulder surgery. In the absence of neuraxial and peripheral nerve blocks, opioid consumption after shoulder surgery has been purported to rival the one recorded for thoracotomy. Interscalene brachial plexus blocks (ISBB) constitute the gold standard for analgesia after shoulder procedures. Compared with parenteral opioids, ISBB results in lower pain scores improved patient satisfaction [4]. ISBB is highly utilized in clinical practice as it provides anesthesia and analgesia to the shoulder and lateral aspects of the arm and the forearm, reducing opioid consumption and subsequent opioid-related adverse effects [5]. However, ISB is associated with numerous complications and adverse effects3 such as phrenic nerve palsy (100%), recurrent laryngeal nerve block (3 - 21%), stellate ganglion block (5 - 75%) (Horner's syndrome), spinal (0.4 - 4%) and epidural anesthesia (2.2%), and convulsions (0.2 - 3%) at standard volumes of 20 - 30 ml. Phrenic nerve block is associated with significant reductions in ventilatory function including a 21 - 34% decrease in forced vital capacity (FVC), 17 - 37% decrease in forced expiratory volume, and 15.4% decrease in peak expiratory flow rate. The most common adverse effect after ISB remains the occurrence of ipsilateral phrenic nerve block. Although well tolerated by healthy subjects, HDP becomes a prohibitive risk for patients with pulmonary pathology, who may be unable to withstand the 30% reduction in FVC. Viable diaphragm-sparing alternatives to ISB should achieve three separate and distinct goals: adequate surgical anesthesia (without general anesthesia), adequate postoperative analgesia, and low incidence of HDP. Alternative nerve blocks are performed in shoulder surgery to prevent HDP. Therefore, different approaches such as suprascapular nerve block, costoclavicular block, shoulder block, supraclavicular block, combined infraclavicular and suprascapular block, which are defined as diaphragm sparing blocks, are recommended.

Our study aimed to investigate the minimum effective local anesthetic volume in postoperative analgesia of the anterior suprascapular nerve block (ASSB) and the maximum local anesthetic volume that can be diaphragm-sparing. Our secondary aim is to reveal an important parameter in the diaphragm sparing nerve blocks. The volume of a local anesthetic to be administered should be expected to have a common volume that is the most effective and protects the diaphragm. We envisioned that this should be defined as the minimum target-specific volume (MTsV).

Adults (over 18 years of age) with the American Society of Anesthesiologists Physical Condition classification I to III who are scheduled to undergo unilateral ambulatory arthroscopic shoulder surgery under general anesthesia will be included in the study. Written informed consent will be obtained from all study subjects before participation in this study. Surgical procedures are planned to include shoulder arthroscopy, rotator cuff repair, acromioplasty, Bankart repair, and superior labrum anterior-posterior repair. Patients with a history of serious broncho-pulmonary disease, known phrenic nerve pathology, existing neurological deficits or neuropathy involving the brachial plexus on the surgical side, contraindications to nerve blocks (infection, bleeding diathesis, allergy to local anesthetics), or history will be excluded from the study. A full pre-operative evaluation will be performed with the necessary laboratories the day before the surgery, and written informed consent will be obtained.

The 0.5% initial injected volume of bupivacaine was 10 mL, providing a complete sensory block of anterior suprascapular nerve block based on our clinical experience. According to the Dixon and Massey [10] up-down method, the 0.5% bupivacaine volume used for a given patient was determined by the result of the previous block, as defined above as block success. Once effective ASSB is achieved, the volume of bupivacaine 0.5% to the next patient will be reduced by 1 mL. Conversely, in case of block failure, the volume of 0.5% bupivacaine will be increased by 1 mL in the next patient.

An independent observer will assess ipsilateral hemidiaphragmatic motion by real-time M-mode ultrasonography using a 1 to 5 MHz broadband phased array US probe (Philips CX50). Patients were examined in an upright sitting position and scanned from a low intercostal or subcostal approach using the liver or spleen as the acoustic window. The range of diaphragm movement from the resting expiratory position to deep inspiration (sigh test) and the range of diaphragm movement from the resting expiratory position when quickly inhaling through the nose (sniffing test) will be recorded. More than 75% hemidiaphragmatic movement reduction, no movement, or paradoxical movement will be considered complete paresis. Between 25% and 75%, hemidiaphragmatic movement decrease was considered partial paresis, and less than 25% hemidiaphragmatic movement decrease paresis was considered absent. The movement of the diaphragm will be measured in centimeters. The normal caudal movement was positive (+), paradoxical head movement was negative (-). Each test will be performed three times, and the values will be averaged. All measurements will be made before (beginning) and 30 minutes after the block.

Fifty minutes after the block performance, general anesthesia will be given using a standard protocol of intravenously administered propofol 2 mg/kg, Fentanyl 1 ug/kg, and rocuronium 0.6 mg/kg. Pain scores of the patients will be recorded for 48 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* adults (age greater than 18 yr) with American Society of Anesthesiologists Physical Status classification I to III scheduled to undergo unilateral arthroscopic shoulder surgery under general anesthesia

Exclusion Criteria:

* dementia
* chronic opioid consumption
* chronic pain disease
* chronic obstructive pulmonary disease
* history of serious lung disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age greater than 18 years with American Society of Anesthesiologists Physical Status classification I to III scheduled to undergo unilateral arthroscopic shoulder surgery patients under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
postoperative analgesia | postoperative 48 hours
  minimum effective local anesthetic volume in postoperative analgesia of the anterior suprascapular nerve block (ASSB) and the maximum local anesthetic volume that can be diaphragm-sparing.

SECONDARY OUTCOMES:
diaphragm sparing nerve block | 0 and 30 min after the nerve block
  The volume of local anesthetic to be administered should be expected to have a common volume that is the most effective and protects the diaphragm. We envisioned that this should be defined as the minimum target-specific volume (MTsV).

CONTACTS AND LOCATIONS:
Locations (1):
- Amerikan Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ullah H, Samad K, Khan FA. Continuous interscalene brachial plexus block versus parenteral analgesia for postoperative pain relief after major shoulder surgery. Cochrane Database Syst Rev. 2014 Feb 4;2014(2):CD007080. doi: 10.1002/14651858.CD007080.pub2. PMID 24492959
- [Background] Fredrickson MJ, Krishnan S, Chen CY. Postoperative analgesia for shoulder surgery: a critical appraisal and review of current techniques. Anaesthesia. 2010 Jun;65(6):608-624. doi: 10.1111/j.1365-2044.2009.06231.x. PMID 20565394
- [Background] Abdallah FW, Halpern SH, Aoyama K, Brull R. Will the Real Benefits of Single-Shot Interscalene Block Please Stand Up? A Systematic Review and Meta-Analysis. Anesth Analg. 2015 May;120(5):1114-1129. doi: 10.1213/ANE.0000000000000688. PMID 25822923
- [Background] Kim DH, Lin Y, Beathe JC, Liu J, Oxendine JA, Haskins SC, Ho MC, Wetmore DS, Allen AA, Wilson L, Garnett C, Memtsoudis SG. Superior Trunk Block: A Phrenic-sparing Alternative to the Interscalene Block: A Randomized Controlled Trial. Anesthesiology. 2019 Sep;131(3):521-533. doi: 10.1097/ALN.0000000000002841. PMID 31283740
- [Background] Ilfeld BM, Morey TE, Wright TW, Chidgey LK, Enneking FK. Continuous interscalene brachial plexus block for postoperative pain control at home: a randomized, double-blinded, placebo-controlled study. Anesth Analg. 2003 Apr;96(4):1089-1095. doi: 10.1213/01.ANE.0000049824.51036.EF. PMID 12651666
- [Background] McNaught A, Shastri U, Carmichael N, Awad IT, Columb M, Cheung J, Holtby RM, McCartney CJ. Ultrasound reduces the minimum effective local anaesthetic volume compared with peripheral nerve stimulation for interscalene block. Br J Anaesth. 2011 Jan;106(1):124-30. doi: 10.1093/bja/aeq306. Epub 2010 Nov 8. PMID 21059701
- [Background] Urmey WF, Talts KH, Sharrock NE. One hundred percent incidence of hemidiaphragmatic paresis associated with interscalene brachial plexus anesthesia as diagnosed by ultrasonography. Anesth Analg. 1991 Apr;72(4):498-503. doi: 10.1213/00000539-199104000-00014. PMID 2006740
- [Background] Tran DQ, Elgueta MF, Aliste J, Finlayson RJ. Diaphragm-Sparing Nerve Blocks for Shoulder Surgery. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):32-38. doi: 10.1097/AAP.0000000000000529. PMID 27941477
- See also: Related Info — https://www.scirp.org/(S(351jmbntvnsjt1aadkposzje))/reference/ReferencesPapers.aspx?ReferenceID=1752894